CLINICAL TRIAL: NCT01257360
Title: NEO-RIT - Panitumumab in Combination With Radiotherapy in Patients With Locally Advanced RAS Wildtype Rectal Cancer (Clinical Stages II and III)
Brief Title: Panitumumab in Combination With Radiotherapy in Patients With Locally Advanced RAS Wildtype Rectal Cancer (Clinical Stages II and III)
Acronym: NEO-RIT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: WiSP Wissenschaftlicher Service Pharma GmbH (Other)
Collaborators: Gesellschaft fur Medizinische Innovation - Hamatologie und Onkologie mbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WISP_AG52; 2009-016782-28 (EudraCT Number); GMIHO 009/2009 (Other: GMIHO mbH)
Record Dates: First submitted 2010-12-01; First posted 2010-12-09 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Rectal Cancer
Keywords: RAS-Wildtype; Radiotherapy; Neoadjuvant treatment
MeSH Terms: conditions — Rectal Neoplasms | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Panitumumab — Panitumumab 6 mg/kg BW will be administered IV every 2 weeks (q2w) on day -14, 1, 15, 29 (and 43, in case radiotherapy is still ongoing due to delays) of the radiotherapy.
  Other Names: Vectibix
Radiation: Radiation of the pelvis — Radiation is applied at single doses of 1.8 Gy at the ICRU 50 reference point, once daily, five times a week, adding up to 28 fractions over almost 6 weeks and a total reference dose of 50.4 Gy.

SUMMARY:
The objective of this trial is to obtain evidence that, in patients with RAS wildtype tumors, a chemotherapy-free combined modality treatment with panitumumab is clearly superior to radiotherapy alone and achieves a pCR rate comparable to that after radiochemotherapy including two-drug combinations while reducing the toxicity compared to these two-drug regimens.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of locally advanced rectal cancer (stage II or III) localised 0 - 12 cm ab ano as measured by rigid rectoscopy (i.e. lower and middle third of the rectum)
* Staging requirements: trans-rectal endoscopic ultrasound (EUS) and magnetic resonance imaging (MRI)
* Sufficient representative sample material for RAS analysis
* Wild-type RAS (determined by an accredited local laboratory, if not available by pathology of Mannheim university)

  * RAS wild-type tested in

    * KRAS exon 2 (codons 12/13)
    * KRAS exon 3 (codons 59/61)
    * KRAS exon 4 (codons 117/146)
    * NRAS exon 2 (codons 12/13)
    * NRAS exon 3 (codons 59/61)
    * NRAS exon 4 (codons 117/146)
* Informed consent of the patient
* Aged at least 18 years
* WHO Performance Status 0-2
* Life expectancy of al least 12 weeks
* Adequate haematological, hepatic, renal and metabolic function parameters:

  * Leukocytes > 3000/mm³
  * ANC ≥ 1500/mm³
  * Platelets ≥ 100,000/mm³
  * Hb > 9 g/dl
  * Creatinine clearance ≥ 50 ml/min and serum creatinine ≤ 1.5 x upper limit of normal
  * Bilirubin ≤ 1.5 x upper limit of normal
  * GOT-GPT ≤ 2.5 x upper limit of normal
  * AP ≤ 5 x upper limit of normal
  * Magnesium ≥ lower limit of normal
  * Calcium ≥ lower limit of normal

Exclusion Criteria:

* Lower border of the tumor localised more than 12 cm ab ano as measured by rigid rectoscopy
* Distant metastases (to be excluded by CT scan of the thorax and abdomen)
* cT4 tumor (as determined by MRI and/or endorectal ultrasound)
* Risk of tumor involvement of the circumferential resection margin, according to the MRI assessment
* Sphincter sparing is the major reason for choosing the neoadjuvant treatment approach
* Prior antineoplastic therapy for rectal cancer
* Prior radiotherapy of the pelvic region
* Major surgery within the last 4 weeks prior to inclusion
* Subject pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment
* Subject (male or female) is not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment (adequate: oral contraceptives, intrauterine device or barrier method in conjunction with spermicidal jelly)
* Serious concurrent diseases
* On-treatment participation in a clinical study in the period 30 days prior to inclusion
* Clinically significant cardiovascular disease in (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year before enrolment
* History of interstitial lung disease, e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan
* History of HIV infection
* Prior or concurrent malignancy (≤ 5 years prior to enrolment in study) except non-melanoma skin cancer or cervical carcinoma FIGO stage 0-1 if the patient is continuously disease-free
* Known allergic reactions on study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-12; Primary Completion 2016-01 (Actual); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Rate of pathological complete remissions | 15 weeks (average) after start of treatment (at surgery)
  The rate of pathological complete remissions is determined after tumor resection following neoadjuvant treatment.

SECONDARY OUTCOMES:
Toxicity according to NCI CTCAE
Frequency of surgical morbidity and complications | Within four weeks after surgery
pTNM findings in relation to initial cTNM staging | At surgery
Regression grading according to Dworak | At surgery
Clinical response rates (CR/PR/SD/PD) after neoadjuvant treatment | Before surgery
Correlative biomarker analyses

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Hofheinz, Prof. Dr. med., Principal Investigator — Tagestherapiezentrum am ITM & III. Medizinische Klinik, Universitätsmedizin Mannheim
Locations (5):
- Germany (5):
  - Klinikum Esslingen Klinik für Onkologie, Gastroenterologie und Allgemeine Innere Medizin, Esslingen am Neckar
  - Klinik für Strahlentherapie und Onkologie, Universitätsklinikum Frankfurt am Main, Frankfurt am Main
  - SLK-Kliniken Heilbronn GmbH Medizinische Klinik III, Heilbronn
  - Tagestherapiezentrum am ITM & III. Medizinische Klinik, Universitätsmedizin Mannheim, Mannheim
  - Prosper Hospital Medizinische Klinik I, Recklinghausen